CLINICAL TRIAL: NCT03870919
Title: PALbociclib in Advanced Breast Cancer: Therapy INtegrating locorEgional Treatment and Palbociclib in de Novo, Treatment Naive, Stage IV ER+, HER2- Breast Cancer Patients
Brief Title: Locoregional Treatment and Palbociclib in de Novo, Treatment Naive, Stage IV ER+, HER2- Breast Cancer Patients
Acronym: PALATINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/1814; 2019-A00570-57 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Stage IV; Radiotherapy; Surgery
Keywords: therapies combination
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib + locoregional treatment (Other): All patients will receive the standard of care treatment ie Palbociclib + letrozole for 24-26 weeks (a delay of +/- 2 weeks to initiate the locoregional treatment is authorized after the day 1 of cycle 1 of palbociclib plus letrozole). After this period, patient will have the most adapted locoregional treatment ie surgery (conservative or mastectomy) with or without radiotherapy, or radiotherapy. The palbociclib will be continued until progression
  Interventions: Drug: Palbociclib; Other: locoregional treatment

INTERVENTIONS:
Drug: Palbociclib — The included patients will first receive the following systemic treatment according standard of care:
  * Non-steroidal aromatase inhibitor (letrozole)
  * Palbociclib
  * Monthly Luteinizing hormone-releasing hormone (LHRH) analogue for non-menopausal patients only. Surgical bilateral oophorectomy is an acceptable option.
Other: locoregional treatment — After normally 6 courses of systemic treatment initiation, the loco-regional treatment of the primary tumour will be performed: surgery (conservative or mastectomy) with or without radiotherapy, or radiotherapy

SUMMARY:
Approximately 3.5% to 6% of newly diagnosed breast cancer patients are stage IV metastatic. De novo metastatic breast cancer accounts for 20% to 25% of these cases. Despite a decrease in mortality in Europe and North America due to early detection and access to treatment, breast cancer remains the 2ⁿᵈ leading cause of cancer deaths in developed countries after lung cancer and the world's leading cause.

In the ESME French national retrospective cohort (NCT03275311), the newly diagnosed estrogen receptor (ER)-positive and HER2-negative (luminal) metastatic patients had a 59.1 months overall survival (OS) for pre-menopausal women and 44.7 months for postmenopausal women. In the same cohort, the median OS was 47.4 months for de novo metastatic patients with hormone receptor (HR)-positive / HER2-negative breast cancer.

The most important current treatment for metastatic breast cancer remains systemic therapy. Surgery and radiation are mainly used to treat symptoms. However, more than 15 retrospective studies have assessed the impact of locoregional treatment on relapse and OS. These studies suggested an improvement of the OS in patients with de novo metastatic breast cancer thanks to the addition of locoregional treatment to systemic therapy. Recent data from the ESME cohort suggest that patients with de novo luminal or HER2-positive metastatic breast cancer may benefit from local treatment of the primary tumor.

Several prospective trials have attempted to demonstrate the benefit of locoregional treatment with mixed results. This can be explained by a limited power of statistical analysis, on the recruitment of patients with breast cancer of all types, and on a limited access to effective systemic therapies in some cases and all before the area of anti CD4/6 which is the current standard treatment in patients with HR-positive / HER2-negative luminal metastatic disease.

However, guidelines indicate that a "multimodal approach, including curative locoregional treatments, should be considered". As a result, many clinicians offer locoregional treatment of the primary tumor, especially if there is a good response to the first line of systematic treatment.

Taken together, these data underscore the need for an evaluation of the value of combined therapy - endocrine therapy - CDK4/6 inhibitor and locoregional treatment - in this population of patients with newly diagnosed HR-positive / HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women with newly diagnosed and histologically proven de novo adenocarcinoma of the breast, Any T, any N, with at least one metastatic site measurable and/or non-measurable according to Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 and/or PET Response Criteria in Solid Tumours (PERCIST) v1.0 and/or MD Anderson bone response criteria (MDA criteria). For patients with only bone metastases, at least one lytic and non-irradiated lesion must be present NB: Bilateral breast cancer is allowed only if tumours present similar histological criteria (morphological subtype, ER and HER2 status).
2. Estrogen Receptor (ER)-positive and HER2-negative breast cancer. To be considered as ER-positive, the biopsy of the primary tumour must display at least 10% of cancer cells with positive ER staining. HER2-positive is defined as IHC3+ or FISH/CISH amplified according to 2018 criteria
3. Age ≥18 years
4. Eastern Cooperative Oncology Group (ECOG) ≤2
5. Indication for treatment with palbociclib and letrozole (with or without ovarian suppression)
6. Diagnostic FFPE tumour sample and/or frozen primary breast tumour sample available
7. Women of childbearing potential must have a negative serum or urine pregnancy test done within 14 days before inclusion
8. Patients must agree to use adequate contraception methods for the duration of the study and for within 21 days after completing treatment
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and any protocol-related procedures including absence of co-morbidities preventing surgery and or radiotherapy and any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. Those conditions should be discussed with the patient before registration in the trial
10. Patient affiliated to a social security system
11. Written informed consent obtained prior to performing any protocol-related procedures including screening evaluations

Exclusion Criteria:

1. Patients with advanced, symptomatic, visceral spread at a risk for short-term, life-threatening complications according to investigator judgement and at risk for visceral crisis as defined by ABC4*
2. Women with previously diagnosed and treated ipsilateral adenocarcinoma of the breast
3. Women with previously treated or concomitant contralateral breast cancer except for Ductal carcinoma in situ (DCIS) treated with curative intent
4. Patients with another concomitant cancer
5. Concurrent enrolment in another clinical trial in which investigational therapies are administered or administration of an investigational drug within 30 days before inclusion
6. Pregnant women or women who are breast-feeding
7. Inability or willingness to swallow oral medication
8. HIV, hepatitis (B and C)
9. Active infection
10. Prior therapy for metastatic breast cancer (systemic or local)
11. Persons deprived of their freedom or under guardianship or incapable of giving consent

    * Visceral crisis is defined as severe organ dysfunction as assessed by signs and symptoms, laboratory studies and rapid progression of disease. Visceral crisis is not the mere presence of visceral metastases but implies important visceral compromise leading to a clinical indication for a more rapidly efficacious therapy, particularly since another treatment option at progression will probably not be possible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate in patients receiving the letrozole plus palbociclib combination plus locoregional treatment | 24 months
  Overall survival

SECONDARY OUTCOMES:
Clinical response rate on both primary tumour and metastasis disease | 24 months
  Follow-up of the disease status by imaging exams until surgery
Pathological response rate in primary tumour | 26 weeks
  Pathological response (tumour size, cellularity... ) evaluated at the surgery or at the biopsy
Conversion rate of breast surgery (conservative-radical) | 26 weeks
  Rate of modification of indication of mastectomy
Locoregional control rate | 60 months
  Rate of locoregional recurrence after surgery and/or radiotherapy
Progression-free survival (PFS) | 60 months
  Follow-up of the disease status by imaging exams
Overall survival | 60 months
Incidence of combined therapies in terms of adverse events | 60 months
  Will be evaluated using the National Cancer Institute - common terminology criteria for adverse events (NCI-CTCAE) v5.0
Registration of post letrozole-CDKi therapies | 60 months
  Records of cancer treatments prescribed to patients after disease progression
Evolution of quality of life during treatment | 60 months
  self-administered questionnaire of quality of life EORTC QLQ-C30 taking into account the patient's activity and his/her physical and psychological state
Evolution of quality of life during treatment | 60 months
  self-administered questionnaire of quality of life EORTC QLQ-BR23, complementary module to QLQ C30 questionnaire, is more specifically interested in patients with se cancer and the impact of treatment on their lives
Evolution of quality of life during treatment | 60 months
  self-administered questionnaire of quality of life Euroquol EQ-5D-5L consists of a descriptive system and a visual scale

CONTACTS AND LOCATIONS:
Overall Officials: Claire Bonneau, MD, Principal Investigator — Institut Curie
Locations (26):
- France (26):
  - Institut de Cancérologie de l'Ouest-Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre François Baclesse, Caen
  - Hôpital privé sainte Marie, Chalon-sur-Saône
  - CH Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital St Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital saint Eloi CHU Montpellier, Montpellier
  - ICM Val d'Aurelle, Montpellier
  - Institut Curie Site Paris, Paris
  - Hôpital Saint Louis APHP, Paris
  - Hôpital St Joseph, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier de Pau, Pau
  - CH René Dubos, Pontoise
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie Hôpital René Huguenin, Saint-Cloud
  - Hôpital Privé à Saint Grégoire, Saint-Grégoire
  - GCS RISSA - Institut de cancérologie Paris Nord, Sarcelles
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.